CLINICAL TRIAL: NCT06539728
Title: Validation of Texture-Changing Tactile Coatings for Potential Use in Accessible At-Home Care
Brief Title: Validation of Texture Changing Coatings for Use in At-Home Rapid Tests
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2181777
Record Dates: First submitted 2024-07-10; First posted 2024-08-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-06

CONDITIONS: Vision, Low; Blindness
Keywords: Tactile Aid
MeSH Terms: conditions — Vision, Low; Blindness | interventions — Drug Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interaction with Coated Surfaces (Experimental): Participants in this arm will interact with the device and surface coated with the polymer-antibody coating. Subjects will be trained with a "positive" test and "negative" test prior to device testing. Subjects will then administer the synthetic saliva themselves and asked to determine if there was COVID antigen in the saliva by touching the device to compare the test patch to the positive and negative control patches. Subjects will also rate device usability.
  Interventions: Diagnostic Test: Interaction with Mock COVID-19 Rapid Antigen Test and Reference Surfaces; Diagnostic Test: Biomechanical Measurements; Behavioral: Psychophysical Tasks

INTERVENTIONS:
Diagnostic Test: Interaction with Mock COVID-19 Rapid Antigen Test and Reference Surfaces — Participants will drop a saline solution with proteins onto the testing device. They will wait for it to dry and then report on the tactile sensation and overall feel of the surface. Feedback will include comparisons with the two reference surfaces. The primary goal is to determine the presence of mock COVID antigen in synthetic saliva using the device, which aligns with the goals of diagnostic testing.
Diagnostic Test: Biomechanical Measurements — Participants may have biomechanical measurements recorded, such as placing samples on a scale to measure downward force or using medical tape with a flexible wire to track finger motion. These measurements are likely aimed at objectively assessing how participants interact with the surfaces and their physical responses to tactile stimuli.
Behavioral: Psychophysical Tasks — Participants may alternatively be asked to perform standardized psychophysical tasks, such as Two Alternative Forced Choice tests, Odd-Man Out tests, or Magnitude Estimation tests. These tasks will provide structured comparisons and quantitative data on participants' perception and preferences regarding tactile qualities. The tasks are designed to evaluate participants' perception and preferences regarding tactile qualities, which involves behavioral responses to sensory stimuli.

SUMMARY:
At-home testing is an important part of mitigating the spread of COVID-19, but these tests are not accessible to people with low vision or blindness. Instead of adapting to a technology originally built for sighted people, investigators propose a no-power version that reports test results through a texture change, which people can feel by touch. This platform could be used not only for COVID, but also for other diagnostics, and will promote the independence and privacy for people with low vision or blindness by removing the need for human assistance or an internet connection.

DETAILED DESCRIPTION:
Current at-home COVID tests are not accessible to people with low vision or blindness. To interpret results, people with low vision or blindness may need a sighted assistant, an internet-based image recognition tool, or some other sort of powered implement. Instead of adapting to technologies developed for sighted people, investigators propose a new platform which provides a no-power tactile readout, i.e., a texture change, to interpret test results. Although COVID antigens are at relatively low concentrations in human saliva, by relying on surface chemistry effects, a relatively small amount of sample can be designed to cause a significant texture change. This project will develop a new class of antibody-conjugated polymers which, in a saliva sample, bind to COVID antigen. In conjunction, investigators will also develop a test surface designed to maximize tactile feedback upon antigen binding. Upon binding to the test surface, a COVID positive surface will feel distinctive from the negative control, like distinguishing between plastic and glass. To optimize polymer design and test surface design, investigators use a combination of materials characterization, mechanical testing, human testing, and computational techniques. The project culminates by having low vision or blind users test the device with synthetic saliva solutions containing COVID antigen, present as innocuous protein isolates. Subjects will receive synthetic saliva with and without COVID antigen, and using our platform, will be asked to determine if the synthetic saliva did contain the COVID antigen. As a platform, the technology is not limited to COVID, but could be adapted to either new variants or other use cases, such as pregnancy tests. Investigators expertise combines accessibility experts, synthetic chemists, human psychophysics, computational simulations, surface science, and mechanics. To maximize project success, the project includes people with visual impairments at all stages to ensure practicality.

ELIGIBILITY:
Inclusion Criteria:

* Visual Impairment: Participants should be blind or visually impaired for greater than 10 years, either congenitally or acquired.
* Tactile Aid Usage: Participants must use tactile aids regularly.
* Mathematical Knowledge: Participants should have a basic understanding of mathematical plots, equivalent to at least high school geometry.

Exclusion Criteria:

* Limb Conditions: Participants with amputations or outer extremity conditions affecting hand use will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Success rate of identifying whether the model test is positive or negative | Through study completion, an average of 1 year
  After familiarization, test trials will involve participants dropping a test solution onto the device with a test slab as well as positive and negative control slabs. They will be asked to identify whether the test is positive or negative, based on how the test slab feels to the touch compared to the controls. Participants will be evaluated on whether or not their response is correct. This will be repeated 10 times per participant to record a percentage of success.
Response time of each trial of a participant identifying whether the model test is positive or negative | Through study completion, an average of 1 year
  A Qualtrics form will be used to record participant responses. Each trial will have its own page on the form during data collection. A trial will begin when the test administrator opens its page, and participants will be prompted to decide whether the device is displaying a positive or negative result. Once participants choose, the administrator will select their answers on the form, and the time to the last click will be recorded as their response time. This will be repeated 10 times.
Usability feedback | Through study completion, an average of 1 year
  Subjects participating in the clinical trial will be invited to provide feedback on the usability and their preferences regarding the tactile aid introduced in the study. The assessment will be conducted using a modified Likert scale. This outcome aims to gather subjective experiences related to the use of new tactile aids throughout the trials. Throughout the study, participants will be consistently asked to comment on the usability and their preferences based on the tactile aid. This ongoing feedback will enable a comprehensive understanding of their experiences over time.
  Modified Likert Scale:
  Strongly Disagree Disagree Somewhat Disagree Neutral Somewhat Agree Agree Strongly Agree Extremely Agree Exceptionally Agree
  Title: Usability of Tactile Aid Min: 1 Max: 9 Higher the score, the better the outcome/ usability of the tactile aid.
General feedback | Through study completion, an average of 1 year
  Subjects participating in the clinical trial will be invited to provide feedback on the usability and their preferences regarding the tactile aid introduced in the study. The assessment will be conducted by asking participants for general feedback on the device they used. Throughout the study, participants will be consistently asked to comment on the usability and their preferences based on the tactile aid. This ongoing feedback will enable a comprehensive understanding of their experiences over time.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No